CLINICAL TRIAL: NCT01746615
Title: Assessment of Retinal Vessel Diameters and Red Blood Velocities in Patients With BRVO and Healthy Subjects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Gerhard Garhofer, Assoc. Prof. PD Dr., Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: OPHT-260612
Record Dates: First submitted 2012-12-07; First posted 2012-12-11 (Estimated); Last update posted 2022-04-07 (Actual); Status verified 2022-04

CONDITIONS: Branch Retinal Vein Occlusion; Retinal Blood Flow; Retinal Oxygen Saturation
Keywords: branch retinal vein occlusion; dynamic vessel analyzer; fourier-domain OCT; retinal oxygen saturation
MeSH Terms: conditions — Retinal Vein Occlusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 30 Patients with BRVO in one eye (Experimental)
  Interventions: Device: Dynamic Vessel Analyzer; Other: Bidirectional Fourier-Domain Optical Coherence Tomography (FDOCT)
- 30 healthy age and sex matched controls (Experimental)
  Interventions: Device: Dynamic Vessel Analyzer; Other: Bidirectional Fourier-Domain Optical Coherence Tomography (FDOCT)

INTERVENTIONS:
Device: Dynamic Vessel Analyzer — retinal vessel diameter & oxygen saturation
Other: Bidirectional Fourier-Domain Optical Coherence Tomography (FDOCT) — retinal blood velocity

SUMMARY:
Assessment of retinal vessel calibers combined with bidirectional Fourier domain optical coherence tomography (FDOCT) for measurement of retinal blood velocities is a new and sophisticated method for assessing retinal blood flow in humans. The valid measurement of retinal blood flow is of significant importance, because it is known that major ophthalmic diseases are associated with alterations in blood flow.

As such, retinal vascular occlusive diseases represent a major cause of visual impairment and blindness. The prevalence of the disease is between 0.7 and 1.6%. Compression of the retinal veins at arterio-venous (AV) crossings plays an important role in the development of branch retinal vein occlusion (BRVO). The mechanical narrowing of the vessel lumen is supposed to be the mechanism behind this fact. The present study should elucidate how BRVO influences retinal blood flow at retinal vessel crossings in comparison to healthy control subjects. Retinal blood flow at retinal bifurcations will also be assessed. In addition, a fundus image will be taken to assess retinal oxygen saturation.

For the first time we use a combination of a dynamic vessel analyzer (DVA) with bidirectional Fourier domain optical coherence tomography (FDOCT) to assess retinal blood flow. Whereas the DVA provides information concerning retinal vessel caliber, FDOCT provides laser Doppler information in addition to conventional optical coherence tomography, allowing the observation of blood flow dynamics simultaneously.

In the present study we hypothesize that the DVA in combination with FDOCT is a suitable new tool for the assessment of blood flow in healthy subjects and in patients with BRVO.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for healthy subjects

* Men and women aged over 18 yrs
* Nonsmokers
* Normal findings in the medical history unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 6 Dpt.

Inclusion criteria for patients with BRVO

* Age ≥ 18a
* Patients with branch retinal vein occlusion with a history of 3 to 9 months in one eye
* No history of BRVO in the fellow eye
* Temporal inferior or superior vein occlusion
* Ametropia < 6 Dpt

Exclusion Criteria:

Any of the following will exclude a healthy subject from the study:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study (except oral contraceptive)
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* Blood donation during the previous 3 weeks
* Pregnancy
* Any abnormalities preventing reliable measurements as judged by the investigator

Any of the following will exclude a patient with BRVO from the study:

* Presence of intraocular pathology other than branch retinal vein occlusion
* Blood donation during the previous 3 weeks
* Clinical trial in the 3 week preceding the study
* Pregnancy
* Any abnormalities preventing reliable measurements as judged by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-08 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09-02 (Estimated)

PRIMARY OUTCOMES:
Retinal blood flow | once on the study day

SECONDARY OUTCOMES:
Retinal vessel diameter | once on the study day
Retinal blood velocity | once on the study day
Retinal oxygen saturation | once on the study day

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria